CLINICAL TRIAL: NCT02989636
Title: Phase I Safety Study of Stereotactic Radiosurgery With Concurrent and Adjuvant PD-1 Antibody Nivolumab in Subjects With Recurrent or Advanced Chordoma
Brief Title: Nivolumab With or Without Stereotactic Radiosurgery in Treating Patients With Recurrent, Advanced, or Metastatic Chordoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); Chordoma Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J16138; IRB00117650 (Other: JHM IRB); NCI-2016-01638 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA006973 (NIH); 18-020 (Other: MSKCC); CA209-594 (Other: BMS)
Record Dates: First submitted 2016-12-08; First posted 2016-12-12 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chordoma
MeSH Terms: conditions — Chordoma | interventions — Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (nivolumab) (Experimental): Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 14 days for 8 doses, then every 28 days for a total of 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Arm II (nivolumab, SRS) (Experimental): Patients receive nivolumab as in Arm I. Patients undergo stereotactic radiosurgery (SRS) as per standard of care on day 8 of course 1.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm II (nivolumab, SRS)

SUMMARY:
This phase I trial studies the side effects of nivolumab with or without stereotactic radiosurgery (SRS) in treating patients with chordoma that has come back or spread from where it started to other places in the body. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to normal tissue. It is not yet known whether giving nivolumab with or without stereotactic radiosurgery may work better in treating patients with chordoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety profile of nivolumab alone and nivolumab in combination with stereotactic radiosurgery to treat patients with recurrent or advanced chordoma.

SECONDARY OBJECTIVES:

I. To evaluate toxicity and tolerability of nivolumab alone and nivolumab in combination with stereotactic radiosurgery.

II. To estimate growth modulation index on target lesion. III. To estimate a clinical response (partial response [PR] + complete response [CR] within 6 month + stable disease [SD] beyond 6 months).

IV. To assess progression-free survival and progression-free survival (PFS) rate at 6 months.

V. To assess overall survival rate at 1 year, 3 years and 5 years.

TERTIARY OBJECTIVES:

I. To explore peripheral blood immune response during and after treatment.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 14 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive nivolumab as in Arm I. Patients undergo stereotactic radiosurgery (SRS) as per standard of care on day 8 of course 1.

After completion of study treatment, patients are followed up at 100 days and every 10 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of chordoma; the pathologic confirmation may be from another metastatic site
* Patients may have metastases, with newly identified peripheral metastases
* Cross-sectional imaging evidence of progression of recurrent or metastatic disease
* Previous treatment information (name of agent, treatment starting date, and date of progression) must be available for review
* Measurable disease in one or more site. (Per RECIST criteria: Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 10 mm with CT scan, MRI, or calipers by clinical exam. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters)).
* Karnofsky performance scale >= 70%
* White blood cells (WBC) >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 2 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR according to Johns Hopkins magnetic resonance imaging (MRI) policy
* Women of child bearing potential (WOCBP) should use an adequate method to avoid pregnancy for 5 months plus the time required for nivolumab to undergo approximately five half-lives) after the last dose of investigational drug; in order for a woman to be determined not of child-bearing potential, she must have >= 12 months of non-therapy induced amenorrhea or be surgically sterile
* Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product
* Ability to understand and the willingness to sign written informed consent document(s)

Exclusion Criteria:

* Prior chemotherapy within 21 days or 5 half-lives (whichever is shorter) days of starting treatment
* Prior therapy with investigational drugs within 21 days or at least 5 half-lives (whichever is shorter) before study administration
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PDL-2 antibody
* Neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Known allergy to compounds of similar chemical or biologic composition to nivolumab
* Pregnant or breastfeeding women
* Known history of human immunodeficiency virus
* Active infection requiring therapy, including positive tests for hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA)
* Active autoimmune disease, history of autoimmune disease or history of syndrome that required systemic steroids or immunosuppressive medications, e.g. organ, tissue, or allogenic hematopoietic stem cell transplant (HSCT) recipients. Exceptions include those with resolved childhood asthma/atopy. Subjects with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study. Subjects are also permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Use of any vaccines against infectious diseases (e.g. varicella, influenza, etc.) up to 4 weeks (28 days) before receiving nivolumab
* Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Prior radiation doses equivalent to, or greater than, 8000 cGy in 200 cGy fractions
* Any radiation to the target lesions within 6 months of enrollment
* Unable to meet radiation treatment plan parameters
* Unavailable for follow up visits after treatment
* Prior malignancy unless disease free for ≥ 2 years. Curatively treated basal or squamous cell carcinoma of the skin, totally excised melanoma of stage IIA or lower, low- or intermediate-grade localized prostate cancer (Gleason sum ≤7), and curatively-treated carcinoma in situ of the cervix, breast, or bladder are allowed regardless.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities evaluated according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 12 weeks after initial dose of nivolumab
  Proportion of serious adverse events will be estimated using the binomial distribution along with 95% confidence interval (exact method).

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Kleinberg, MD, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (2):
- United States (2):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No